CLINICAL TRIAL: NCT06909305
Title: Effect of Intraarticular Ozone, Prolotherapy or Dexmedetomidine in Pain Limitation in Knee Osteoarthritis: A Randomized Prospective Study
Brief Title: Effect of Intraarticular Ozone, Prolotherapy or Dexmedetomidine in Pain Limitation in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ghada Abd El-Wahab Saif El-Dien, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Management, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35148/12/21
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Intraarticular; Ozone; Prolotherapy; Dexmedetomidine; Pain; Knee Osteoarthritis
MeSH Terms: conditions — Pain; Osteoarthritis, Knee | interventions — Ozone; Dexmedetomidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ozone group (Experimental): Patients received intraarticular ozone injection.
  Interventions: Drug: Ozone
- Dextrose prolotherapy group (Experimental): Patients received intraarticular dextrose prolotherapy injection.
  Interventions: Drug: Dextrose prolotherapy
- Dexmedetomidine group (Experimental): Patients received intraarticular dexmedetomidine injection.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ozone — Patients received intraarticular ozone injection.
  Arms: Ozone group
Drug: Dextrose prolotherapy — Patients received intraarticular dextrose prolotherapy injection.
  Arms: Dextrose prolotherapy group
Drug: Dexmedetomidine — Patients received intraarticular dexmedetomidine injection.
  Arms: Dexmedetomidine group

SUMMARY:
This study aimed to compare intraarticular ozone injection, prolotherapy, or dexmedetomidine effectiveness in knee osteoarthritis patients.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a heterogeneous group of disorders of different etiologies with similar biological, morphological, and clinical manifestations and outcomes. The intraarticular injection has been recommended to alleviate the pain in the knee joint.

Ozone therapy has long been used in the management of OA. Furthermore, it has been shown to not cause a significant inflammation process or cartilage degradation. Prolotherapy is a procedure where a natural irritant is injected into the soft tissue of an injured joint. Dexmedetomidine is a selective α2-adrenergic agonist with considerable sedative and analgesic actions.

ELIGIBILITY:
Inclusion Criteria:

* Age from 30 to 65 years.
* Both genders.
* Patients diagnosed with stage 1-3 osteoarthritis according to the Kellgren-Lawrence Classification System (K-L).

Exclusion Criteria:

* Patient refusal.
* History of knee trauma within the past month.
* Rheumatic disease.
* Pregnancy.
* Any surgical intervention of the knee.
* Severe cardiovascular disease.
* Morbid obese patients (body mass index (BMI) of >35 kg/m2).
* Local infection at the site of injection.
* Bleeding diathesis.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Analgesic requirement | 3 months after the procedure
  Analgesic requirements for pain control after injection were recorded.

SECONDARY OUTCOMES:
Improvement of lifestyle | 3 months after the procedure
  Improvement of lifestyle was assessed using the Western Ontario Mac Master Osteoarthritis Index (WOMAC-OI) scale. The Likert type of the WOMAC Persian version was employed in this paper. The Persian version is a dependable and uncomplicated procedure that provides five responses: extreme (4), severe (3), moderate (2), mild (1), and none (0). The patients' stiffness, pain, and functional restriction are all represented by the higher scores.
Improvement of knee joint cartilage regeneration | 3 months after the procedure
  Improvement of knee joint cartilage regeneration was assessed using the Kellgren-Lawrence Classification System (K-L). K-L: which categorize knee OA into four stages based on radiological findings: Grade 4 (severe): Marked joint space narrowing, large osteophytes, severe sclerosis, and definite deformity of bone ends. Grade 3 (moderate): Moderate multiple osteophytes, some sclerosis, definite joint space narrowing, and potential deformity of bone ends. Grade 2 (minimal): Definite osteophytes and potential joint space narrowing. Grade 1 (doubtful): Possible osteophytic lipping and doubtful joint space narrowing.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.